CLINICAL TRIAL: NCT01368120
Title: Antimicrobial Activity of IV Clear™ Dressing - Prevention of Antimicrobial Regrowth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Covalon Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TP-014
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Skin Flora Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV Clear™ (Experimental)
  Interventions: Device: IV Clear™ Dressing
- Tegaderm CHG™ (Active Comparator)
  Interventions: Device: Tegaderm CHG™
- Vehicle Control Dressing (Placebo Comparator)
  Interventions: Device: Silicone Vehicle Control Dressing

INTERVENTIONS:
Device: IV Clear™ Dressing — Polyurethane film, silicone adhesive dressing with chlorhexidine and silver
  Arms: IV Clear™
Device: Tegaderm CHG™ — Polyurethane film, polyacrylate adhesive and a polyol hydrogel containing 2% w/w chlorhexidine gluconate
  Arms: Tegaderm CHG™
Device: Silicone Vehicle Control Dressing — Polyurethane film with silicone adhesive dressing, without antimicrobials
  Arms: Vehicle Control Dressing

SUMMARY:
The purpose of this study is to assess the surface cutaneous antimicrobial activity of IV Clear™ Dressing, Tegaderm CHG™ Dressing and a Silicone Vehicle Control Dressing.

DETAILED DESCRIPTION:
A single center, within-subject randomized study design in healthy adult subjects with a history of high bacteria counts on their upper back, meeting the inclusion criteria.

Antimicrobial efficacy will be measured by determining the mean number of Colony Forming Units (CFUs) per square centimetre (cm²) of skin prior to treatment (baseline measurement), following preparation with 70% isopropyl alcohol, and following post treatment samples.

The goal of this study is to demonstrate that IV Clear™ is as effective as or better than Tegaderm™ CHG dressing in preventing regrowth of cutaneous microbial flora on test subjects.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years of age and ≤ 65 years of age
* Are in good health, as evidenced by response to the demographics/dermatological medical history form
* Are willing to refrain from using antimicrobial soaps for bathing and showering during the entire study
* Are willing to refrain from swimming in chemically treated pool or hot tub for duration of study
* Are willing to refrain from using antimicrobial/medicated lotions and creams for duration of study, unless prescribed by a physician for an intercurrent illness
* Are willing to refrain from using topical or systemic antibiotic medication for duration of study, unless prescribed by a physician for an intercurrent illness
* Are willing to refrain from use of body powders and fabric softeners
* Are willing to use soap and shampoo and antiperspirant/deodorant provided exclusively during study
* Have qualification screening bacterial counts of ≥ 2.5 log10 CFU/cm² on two contralateral sites on the upper back
* Are willing to comply with all study protocol requirements

Exclusion Criteria:

Subjects will not be enrolled in the study if they:

* Are currently pregnant or lactating
* Have been exposed to topical or systemic antimicrobials during two weeks proceeding treatment. This restriction will include, but is not limited to shampoos, lotions, soaps, body powders, and materials such as solvents, acids, or alkalis
* Have known soap, detergent, antibiotic and/or perfume allergies
* Have been medically diagnosed as having a medical condition that precludes participation, such as: diabetes, hepatitis, an organ transplant, a medical surgical implant or an immune compromised system
* Have any medical condition which in the opinion of the Investigator prelude participation
* Have swam in chemically treated pools or hot tubs two weeks prior to any microbial sampling
* Have used UV tanning lamps two weeks prior to any microbial sampling
* Have tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders on test sites
* Have bathed or showered less than 48 hours prior to any microbial sampling
* Have known sensitivity to adhesive products, or to materials used in test articles
* Have participated in any type of back wash study within 7 days prior to study
* Have a known sensitivity to latex products
* Are not willing to fulfill the requirements of the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in skin microbial colonization over 7-day period of antimicrobial dressing application | Assessed after 4 days and 7 days of dressing application
  Mean number of Colony Forming Units (CFUs) per square centimetre (cm²) of skin prior to treatment (baseline), following prepping with 70% isopropyl alcohol and following post treatment samplings of IV Clear™, Tegaderm™ CHG and Silicone control dressings collected.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Ward, D.O., Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, Miamiville, Ohio, United States